CLINICAL TRIAL: NCT07126132
Title: The Hemopexin-Apolipoprotein B Product: A Novel Biomarker Integrating Oxidative Stress and Lipid Metabolism for Coronary Artery Disease Risk Stratification
Brief Title: Hpx•apoB Product as a Biomarker for Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Shiyan City Renmin Hospital (Other Government)
Responsible Party: Principal Investigator, Qunxiong Fan, Principal investigator, Shiyan City Renmin Hospital
Other Study IDs: syrmyy2018-079
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Fasting blood samples were collected into EDTA-containing tubes. Plasma was separated and used to measure hemopexin (Hpx), apolipoprotein B (apoB), lipid profile, hs-CRP, and other standard laboratory parameters.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary Artery Disease (CAD) Group (n=350): Patients with angiographically confirmed stenosis of ≥50% in at least one major epicardial artery.
  Interventions: Procedure: Coronary Angiography; Diagnostic Test: Hpx•apoB Product Measurement
- Control Group (n=110): Subjects who underwent coronary angiography for symptoms such as chest pain but were found to have no significant coronary stenosis (<50%).
  Interventions: Procedure: Coronary Angiography; Diagnostic Test: Hpx•apoB Product Measurement

INTERVENTIONS:
Procedure: Coronary Angiography — Standard coronary angiography was performed via the radial or femoral approach on all participants to assess the presence and severity of coronary artery disease. Angiograms were used to determine coronary stenosis, which formed the basis for classifying participants into the CAD group (≥50% stenosis) or the control group (<50% stenosis).
Diagnostic Test: Hpx•apoB Product Measurement — Fasting blood samples were collected from all participants to measure the novel Hpx•apoB product. Plasma hemopexin (Hpx) was quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS) and apolipoprotein B (apoB) was measured using standard automated methods. This biomarker was the primary variable of interest for its association with CAD.

SUMMARY:
This was a single-center, cross-sectional study designed to investigate a novel composite biomarker, the Hemopexin-Apolipoprotein B (Hpx•apoB) product, for its association with coronary artery disease (CAD). The study aimed to determine if the Hpx•apoB product could serve as an independent predictor for the presence and severity of CAD and to evaluate its incremental value in improving risk stratification when added to existing clinical risk models.

DETAILED DESCRIPTION:
The pathophysiology of coronary artery disease (CAD) involves complex interactions between lipid dysregulation and oxidative stress. This study proposed and evaluated a novel composite biomarker, the Hemopexin-Apolipoprotein B (Hpx•apoB) product, which integrates a marker of atherogenic particle burden (apoB) with a marker reflecting the systemic response to heme-induced oxidative stress (Hpx). From January 2019 to December 2023, a total of 460 participants were enrolled: 350 patients with angiographically confirmed CAD (≥50% stenosis in a major coronary artery) and 110 control subjects without significant stenosis. Plasma Hpx was quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS). The study used multivariate logistic regression to assess the independent association between the Hpx•apoB product and CAD. Furthermore, its incremental diagnostic value was evaluated by calculating the area under the receiver operating characteristic curve (AUC), net reclassification improvement (NRI), and integrated discrimination improvement (IDI) when added to conventional risk factors and established risk scores (Framingham Risk Score and SCORE2).

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Referred for coronary angiography due to suspected or known CAD.
* Provided written informed consent.

Exclusion Criteria:

* Acute infectious or systemic inflammatory diseases.
* Severe hepatic or renal dysfunction (eGFR < 30 mL/min/1.73m²).
* Malignancy.
* Autoimmune disease.
* A history of major surgery within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of consecutive patients aged 18 years or older who were referred for coronary angiography at the Department of Cardiovascular Medicine, Renmin Hospital, Hubei University of Medicine, due to suspected or known coronary artery disease (CAD). From this population, 460 participants were enrolled after applying inclusion and exclusion criteria. Participants were then allocated into a CAD group (n=350) or a control group (n=110) based on angiographic findings.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Odds Ratio for the Presence of Coronary Artery Disease per Unit Increase in Hpx•apoB Product | Baseline
  This outcome assesses the strength of association between the biomarker and CAD. The plasma concentration of the Hpx•apoB product (Unit: mg²/L²) was used as a continuous variable in a multivariable logistic regression model to predict the presence of CAD. The result is expressed as an Odds Ratio (OR), a unitless measure, with a 95% confidence interval.
Change in Area Under the Receiver Operating Characteristic Curve (AUC) | Baseline
  This outcome measures the incremental predictive value of the Hpx•apoB product. The AUC of a baseline risk model (containing hs-CRP and LDL-C) was compared to the AUC of the same model with the Hpx•apoB product added. The change in AUC (ΔAUC) quantifies the improvement in model discrimination. AUC is a unitless value ranging from 0.5 to 1.0.

SECONDARY OUTCOMES:
Comparison of Hpx•apoB Product Concentration by Number of Diseased Vessels | Baseline
  To assess the association with CAD severity, the mean plasma concentration of the Hpx•apoB product (Unit: mg²/L²) was compared across patient groups categorized by the number of diseased coronary vessels (one-, two-, or three-vessel disease), evaluated using a test for trend.
Correlation Between Hpx•apoB Product and Gensini Score | Baseline
  To assess the association with angiographic severity of CAD, the Spearman correlation coefficient was calculated between the plasma concentration of the Hpx•apoB product (Unit: mg²/L²) and the Gensini score. The Gensini score is a unitless index of atherosclerosis severity.
Correlation Between Hpx•apoB Product and High-Sensitivity C-Reactive Protein (hs-CRP) | Baseline
  The Spearman correlation coefficient was calculated to assess the relationship between the plasma concentration of the Hpx•apoB product and hs-CRP (Unit: mg/L). The correlation coefficient is a unitless value.
Correlation Between Hpx•apoB Product and Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline
  The Spearman correlation coefficient was calculated to assess the relationship between the plasma concentration of the Hpx•apoB product and LDL-C (Unit: mmol/L). The correlation coefficient is a unitless value.
Correlation Between Hpx•apoB Product and Triglycerides (TG) | Baseline
  The Spearman correlation coefficient was calculated to assess the relationship between the plasma concentration of the Hpx•apoB product and triglycerides (Unit: mmol/L). The correlation coefficient is a unitless value.
Correlation Between Hpx•apoB Product and Estimated Glomerular Filtration Rate (eGFR) | Baseline
  The Spearman correlation coefficient was calculated to assess the relationship between the plasma concentration of the Hpx•apoB product and eGFR (Unit: mL/min/1.73m²). The correlation coefficient is a unitless value.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital, Hubei University of Medicine, Shiyan, Hubei, China